CLINICAL TRIAL: NCT00991835
Title: Prospective Multicenter Study to Investigate the Relationship Between the Characteristics of Coronary Artery Plaques and Cardiovascular Events Using Multidetector Computed Tomography Coronary Angiography
Brief Title: Plaque Registration and Event Detection In Computed Tomography
Acronym: PREDICT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, Yasuki Kihara, Department of Cardiovascular Medicine, Graduate School of Biomedical Sciences, Hiroshima University
Other Study IDs: PREDICT2009
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Coronary Artery Disease
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Disruption of an atherosclerotic plaque is responsible for at least two-thirds of acute coronary syndrome. Thus, identification of plaques vulnerable to rupture has become important. The natural history of individual plaques is unknown and needs to be established. Multidetector computed tomography (MDCT) angiography is a useful noninvasive imaging modality for assessing coronary plaque characteristics. Using MDCT, the researchers prospectively investigate the relationship between the characterization of coronary plaques and cardiovascular events in a large multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* patients with known or suspected coronary artery disease.

Exclusion Criteria:

* irregular heart beat,
* known allergy towards the contrast agent,
* renal dysfunction,
* uncontrolled heart failure,
* previous coronary bypass surgery, or pacemaker or ICD implantation, ST elevation MI or unstable hemodynamic condition,
* impossible breath-hold, OR
* end-stage cancer.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients reffered to cardiovascular hospital
Sampling Method: Probability Sample
Enrollment: 3015 (Actual)
Dates: Start 2009-10; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Major cardiac events (Cardiac death and acute coronary syndrome) | 2 years after the CT-scan
All-cause death | 2 years after the CT-scan

SECONDARY OUTCOMES:
All coronary events (Cardiac death, non-fatal MI, unstable angina requiring hospitalization, late coronary revascularizations) | 2 years after CT-scan
All cardiovascular events (Death, acute coronary syndrome, heart failure, cerebral disease, peripheral artery disease, aortic disease, and renal failure) | 2 years after the CT-scan

OTHER OUTCOMES:
Coronary plaque progression and managements for serum cholesterol, blood glucose, renal function and blood pressure: Especially impacts of statin on the changes in coronary plaque characteristics | 2 years after CT

CONTACTS AND LOCATIONS:
Overall Officials: Yasuki Kihara, MD,PhD, Study Chair — Hiroshima University
Locations (1):
- Hiroshima University Graduate School of Biomedical and Health Sciences, Department of Cardiovascular Medicine, Hiroshima, Hiroshima, Japan

REFERENCES:
- [Derived] Yamamoto H, Awai K, Kuribayashi S, Kihara Y; PREDICT Investigators. Rationale and design of the PREDICT (Plaque Registration and Evaluation Detected In Computed Tomography) registry. J Cardiovasc Comput Tomogr. 2014 Mar-Apr;8(2):90-6. doi: 10.1016/j.jcct.2013.12.004. Epub 2014 Jan 8. PMID 24661823